CLINICAL TRIAL: NCT00837720
Title: A 12-Week Open-Label Non-Interventional Evaluation of Atacand® (Candesartan) Efficacy, Tolerability, Compliance and Treatment Satisfaction in Patients With Arterial Hypertension
Brief Title: Evaluation of Atacand® (Candesartan) in Daily Medical Practice
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Meta Jeras, Mr Ph, Regulatory and Medical Affairs Manager, AstraZeneca
Other Study IDs: NIS-CSI-ATA-2005/1
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure; Atacand®; candesartan
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This open label, non-interventional study is to show the efficacy of antihypertensive treatment with Atacand in hypertensive patients. Efficacy is to be evaluated based on the difference in systolic and diastolic blood pressure at baseline and at both follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* a patient with arterial hypertension who has been prescribed Atacand according to physician's judgement, irrespective of the inclusion in the study

Exclusion Criteria:

* hypersensitivity to candesartan or any other ingredient of Atacand
* liver function impairment and/or cholestasis
* severe renal insufficiency
* woman of child-bearing potential and not using appropriate contraceptive measures, pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients (outpatient or hospitalised) in whom Atacand is indicated according to the current Summary of product characteristics (SPC)
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2006-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure reduction | 12 weeks

SECONDARY OUTCOMES:
Incidence and reasons of treatment discontinuation | 12 weeks
Patient treatment satisfaction (using 5-point answering scale) as the measure of the patient's overall tolerance | 12 weeks
Physician overall evaluation of the therapy (using 5-point answering scale) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rok Accetto, MD, Principal Investigator — University Medical Centre Ljubljana